CLINICAL TRIAL: NCT02011828
Title: Ergocalciferol Therapy in Calcidiol Deficient, Hemodialysis Patients on Therapeutic Doses of Paricalcitol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Srinvasan Beddhu, MD, Associate Professor of Medicine, University of Utah
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB_00032685
Record Dates: First submitted 2012-06-13; First posted 2013-12-13 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Inflammation; Insulin Resistance
Keywords: Hemodialysis, paricalcitol
MeSH Terms: conditions — Inflammation; Insulin Resistance | interventions — Ergocalciferols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ergocalciferol, then Placebo (Experimental): Participants first receive Ergocalciferol 50,000 international units (IU)/week for the first 12 weeks. After a 4 week wash-out period, they then receive matching placebo treatment for 12 weeks.
  Interventions: Drug: Ergocalciferol; Drug: Placebo
- Placebo, then Ergocalciferol (Experimental): Participants first receive placebo treatment (matching ergocalciferol 50,000 IU/week) for the first 12 weeks. After a 4 week wash-out period, they then receive ergocalciferol 50,000 IU/week treatment for 12 weeks.
  Interventions: Drug: Ergocalciferol; Drug: Placebo

INTERVENTIONS:
Drug: Ergocalciferol — 50,000 IU/week
Drug: Placebo — Placebo tablet

SUMMARY:
The objective of this study is to determine the effects of cholecalciferol treatment on inflammation and insulin resistance, in patients on hemodialysis that are previously treated with paricalcitol.

Cholecalciferol is produced by the action of sunlight on a cholesterol precursor in the skin. This compound is then converted to calcidiol (25(OH) D3) in the liver, whereupon calcidiol is converted in the kidney to calcitriol (1,25(OH)2D3), the active form of vitamin D. However, recently it has been shown that deficiency of either calcidiol or calcitriol is associated with inflammation, insulin resistance and increased mortality in the general population. Furthermore, when both calcidiol and calcitriol were deficient, the mortality risk was much higher than the deficiency of either alone. A possible explanation is that some of the non-renal tissues might critically depend on the endogenous conversion of calcidiol to calcitriol and not on circulating levels of calcitriol. Thus, low circulating levels of calcidiol might be associated with tissue level functional calcitriol deficiency despite adequate circulating levels of calcitriol.

Therefore, the hypothesis is that:

1. In non-diabetic hemodialysis (HD) patients treated with therapeutic doses of paricalcitol (an analog of calcitriol), calcidiol deficiency is associated with inflammation and insulin resistance and
2. In calcidiol deficient, non-diabetic HD patients with inflammation and treated with therapeutic doses of paricalcitol, cholecalciferol will reverse the calcidiol deficiency and thereby, reduce inflammation and insulin resistance.

Interleulin-6 (IL-6) is thought to play a central role in insulin resistance by down-regulating glucose transporter-4 messenger RNA. Furthermore, IL-6 levels are significantly negatively associated with calcidiol levels, therefore will be measured as the primary outcome.

ELIGIBILITY:
Non-diabetic in-center HD patients on stable doses of paricalcitol over past three months with intact parathyroid hormone (iPTH) in the therapeutic range (150-300 pg/ml) will be identified from review of the dialysis program electronic medical records. Woman in the reproductive age group (ages 18-55), excluding those women who have undergone hysterectomy, oopherectomy will undergo a serum β-HCG levels during the selection process. If β-HCG levels are positive these patients will be excluded from the study.

Inclusion criteria:

* Non diabetic patients on HD, on stable dose of paricalcitol supplements for at least 3 months with iPTH in target range. Of the 60 patients enrolled in the observational component, those with high CRP (> 3 mg/dl) and calcidiol deficiency (< 15 ng/ml) will be eligible to participate in the interventional study.
* As the median CRP in the HEMO Study was 11 mg/L and > 80% of HD patients are calcidiol deficient [10], most of the screened patients will be eligible. In each year, the first 12 patients who meet the above criteria and consent for the interventional component, a randomized cross-over trial of cholecalciferol 50,000 IU/ week vs. matching placebo will be conducted.

Exclusion criteria:

* Diabetic patients, not on paricalcitol, enrolled in other interventional studies, hospitalized in the past month or treated for an infection in the past month and pregnancy.
* We will conduct a pregnancy test for women in the reproductive age group (18-55 years) during the initial screening process. We will obtain serum β-HCG levels to rule out pregnancy and the test will be paid for by the study. The results will be reviewed by the PI. If β-HCG levels are positive these patients will be withdrawn from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of Interleukin-6 (IL-6) | 28 weeks
  Comparison of IL-6 levels after treatment with ergocalciferol and after treatment with placebo

CONTACTS AND LOCATIONS:
Overall Officials: Srinivasan Beddhu, MD, Principal Investigator — University of Utah; Vidya Raj Krishnamurthy, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States